CLINICAL TRIAL: NCT00229645
Title: A Double Blind, Randomized Placebo Controlled Study of the Efficacy, Safety and Tolerability of Immediate-Release Formulation of Quetiapine Fumarate as Potentiation of Selective Serotonin Reuptake Inhibitors, and Serotonin Norepinephrine Reuptake Inhibitors Treatment in Major Depression With Comorbid Anxiety Symptoms
Brief Title: A Double Blind, Randomized Placebo Controlled Study of the Efficacy, Safety and of Quetiapine Fumarate (Seroquel®) as Potentiation SSRI's, and SNRI's Treatment in Major Depression With Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Alexander McIntyre Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1441C00017
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Major Depression With Comorbid Anxiety Symptoms
Keywords: Major Depression; Anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine Fumarate (Seroquel®)

SUMMARY:
Major depression occurs with generalized anxiety disorder and panic disorder in up to 60% of psychiatric and primary care patients.(1) An estimated 85% of adults with depression experience significant symptoms of anxiety and 58% have a diagnosable anxiety disorder during their lifetime.(2) Numerous studies have shown that symptoms of anxiety are frequent in patients with major depressive disorder, and the presence of anxiety symptoms is associated with a more severe and chronic course.(3,4) This comorbidity has been associated with a greater severity of depression, poorer psychosocial functioning, poorer treatment response and higher risk for suicide.

The data suggests that novel antipsychotics have antidepressant and anxiolytic effects. This study will explore the impact of this effect in patients with major depression and comorbid anxiety symptoms.

This study offers the possibility of systematically reviewing the role of quetiapine in depression with anxiety. If the combination of an SSRI or SNRI and quetiapine proves to effective it could offer a viable alternative to widespread benzodiazepine use.

DETAILED DESCRIPTION:
This is a double blind study where patients will be involved and be under treatment for a period of 8 weeks. The initial evaluation will include rating scales measuring depression, anxiety, severity of illness, overall functioning, pregnancy test and clinical evaluations. Patients being treated with a SSRI or SNRI for at least 6 weeks, at therapeutic doses (see table 1.), who still have a HAM-D score of 18 or more, will be randomly assigned to treatment, either with Quetiapine, or Placebo. Patients in the active group will be titrated on a fixed schedule of 50 mg at night for 7 days, 100 mg at night for 7 days, then 200 mg at night for 7 days. After this the dose will be titrated upwards to a maximum of 600mg at night at the discretion of the investigator, using patient tolerance and response as guidelines over the duration of the trial. 200mg is in the range of the average dose in large trials of naturalistic clinical use of quetiapine and is actually much slower than the titration schedule on the package label. Patients that can not tolerate 200mg/day will be withdrawn from the study. Patients should have tried a minimum of 400mg /day before being withdrawn because of lack of efficacy. This dose will remain steady until week 8. Rating scales will be repeated every week during the first 2 weeks, and every 2 weeks up to the end of the study at week 8.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with a DSM IV diagnosis of major depression. 2. Patients will not be on an antipsychotic or a benzodiazepine for at least 7 days prior to entering the study.

  3. Patients will be able to give informed consent. 4. Patients will be male or female between the ages of 18 and 65. 5. Subjects have been treated for at least 6 weeks of single agent SSRI or SNRI therapy at an acceptable dose (see table 1 for detail) in the current episode.

  6. Patients who score at least 18 on the 17-item HAM-D scale, a score of at least 14 on the 14-item HAM-A scale and at least 4 (i.e., moderately ill) on the Clinical Global Impression (CGI) severity scale. Both criteria have to be met at screening and baseline (Study Day 0).

Exclusion Criteria:

* 1. Patients who, in the investigator's opinion, pose a risk for suicide. 2. Present DSM IV diagnosis of substance abuse or dependence within 6 months of the screening visit.

  3. Female subjects of child bearing potential without adequate contraception. Adequate methods of contraception include hormonal contraceptives e.g. oral contraceptives or long term injectable or implantable hormonal contraceptive; double barrier methods, for example condom and diaphragm, condom and foam, condom and sponge; intrauterine device and tubal ligation.

  4. Pregnant or breastfeeding females. 5. Documented disease of the central nervous system including but not limited to stroke, tumor, seizure disorder requiring anticonvulsants, history of brain trauma, chronic infection or a dementing illness.

  6. Hepatic, renal or gastrointestinal disease of sufficient degree to interfere with the excretion, absorption and/or metabolism of trial medication.

  7. Acute, unstable or significant and untreated medical illness. 8. Subjects with narrow angle glaucoma, chronic urinary retention and/or clinically significant prostatic hypertrophy, paralytic ileus or related conditions.

  9. A history of severe drug allergy or hypersensitivity. 10. The use of any of the following potent cytochrome P450 inhibitors in the 14 days preceding randomization (e.g. ketoconazole, itraconazole, fluconazole, erythromycin, troleandomycin clarithromycin, indinavir, nelfinavir, ritonavir and saquinavir).

  11. The use of potent cytochrome P450 inducers (e.g. phenytoin, carbamazepine, barbiturates, rifampin and glucocorticoids) in the 14 days preceding randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-11; Study Completion 2005-04

PRIMARY OUTCOMES:
To compare the efficacy of quetiapine versus placebo over 8 weeks as an adjunctive agent for unipolar non-psychotic adult outpatients on SSRI or SNRI therapy with residual symptoms of depression and comorbid anxiety symptoms. This will be measured by the
1. Hamilton Depression Scale (HAM-D) total score,
2. Hamilton Anxiety Scale (HAM-A) total score

CONTACTS AND LOCATIONS:
Overall Officials: Alexander W McIntyre, FRCPC, Principal Investigator — Dr Alexander McIntyre Inc.
Locations (1):
- Dr. A. McIntyre, Penticton, British Columbia, Canada